CLINICAL TRIAL: NCT03207061
Title: Can 3D Ultrasound be Used as an Alternative to MRI to Assess Myometrial Invasion in Endometrial Cancer?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16HH3687 3D Ultrasound EC
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Endometrial Cancer; Endometrial Neoplasms; Endometrial Hyperplasia
Keywords: endometrial cancer; staging; 3 Dimensional; Ultrasound; Myometrial invasion
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D ultrasound and MRI (Other): All patients with confirmed endometrial cancer will recieve the gold standard pre-operative imaging (MRI) but will also be offered 3D ultrasound.
  Interventions: Diagnostic Test: 3D Ultrasound

INTERVENTIONS:
Diagnostic Test: 3D Ultrasound — A 3D ultrasound will be performed for all patients presenting to the clinic for suspected endometrial cancer (in addition to routine standard of care)

SUMMARY:
Aim: Assess the diagnostic accuracy of 3D Ultrasound, compared to MRI and final histology with respect to myometrial invasion of endometrial cancer.

This study will assess whether 3D ultrasound is accurate at predicting myometrial invasion aqnd lymph node metastasis of endometrial cancer. All patients will receive routine standard of care (MRI). The results of the 3D ultrasound will be compared to the MRI report and final histology.

DETAILED DESCRIPTION:
Aim:

Assess the diagnostic accuracy of 3D Ultrasound, compared to MRI and final histology with respect to myometrial invasion of endometrial cancer.

Background:

When a diagnosis of endometrial cancer is confirmed on biopsy, women get staged to assess the level of spread. Current gold standard is an MRI. A proportion of women, are unable to undergo or complete an MRI scan due to their morbid obesity or claustrophobia. To this end, many have assessed the role of ultrasound in staging endometrial cancer as a cheaper and easier alternative to an MRI. In the last 20 years there has been a rise in the use of 3D ultrasound as it has become commercially available. There is, however a paucity of data on the role of 3D ultrasound in the assessment of myometrial invasion and lymph node metastasis. This research project will assess whether 3D ultrasound is a safe, effective alternative to MRI to assess the depth of spread of womb cancer.

The study:

All women with suspected endometrial cancer will receive a pelvic (internal) ultrasound as per routine care. In addition to the normal 2D ultrasound, women will receive a 3D ultasound and images will be saved. This adds an additional 1-2 minutes scan time.

In those women with confirmed cancer on histology an MRI is performed to assess stage of cancer (current routine standard of care). This will include T1, T2, DWI and contrast enhanced sequences. Patients referred to Hammersmith Hospital from other trusts will also be able to undergo a 3D ultrasound if this was not already performed. Definitive management of endometrial cancer includes a hysterectomy and the surgical specimen will be examined for depth of myometrial invasion and lymph node involved (if removed). In the meantime, the saved 3D ultrasound images will be analysed and rendered to predict the stage of the endometrial cancer and lymph node involvement. The results of 3D ultrasound, and MRI will be compared against the stage found on the gold standard test (on histological examination).

ELIGIBILITY:
Inclusion Criteria:

All women presenting to rapid access gynaecology clinic with postmenopausal bleeding or intermenstrual bleeding or referred with a confirmed diagnosis of endometrial cancer.

Exclusion criteria:

Anyone lacking capacity. <18years old. Pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study looking at endometrial cancer
Enrollment: 500 (Estimated)
Dates: Start 2017-06-13 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of diagnosing myometrial invasion in 3D USS compared to MRI | 1.5 years
  Sensitivity, specificity, negative and positive predictive value in diagnosing myometrial invasion.
Accuracy of predicting lymph node metastasis using 3D USS | 1.5 years
  Measuring 3D volume of tumour and assess if correlation with lymph node metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Charlotte and Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided